CLINICAL TRIAL: NCT01580540
Title: Comparison of the Performance of the Epi proColon and Fecal ImmunochemicalTest Post Colonoscopy in Subjects With Colorectal Cancer and Pre Colonoscopy in Subjects From a Guideline-Eligible Screening Population
Brief Title: Head to Head Study Epi proColon and FIT
Status: Completed | Type: Observational
Sponsor: Epigenomics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Epigenomics-SPR 0022
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A, subjects with colorectal cancer: Subjects between ages 50 and 84 identified to have CRC. Blood and stool specimens are collected and tested after colonoscopy and prior to surgery or other interventions.
- Group B, subjects without CRC: Subjects between ages 50 and 84 who provide stool and blood specimens prior to colonoscopy.

SUMMARY:
The study aims to show non-inferiority in the clinical performance of the investigational assay, Epi proColon, to FIT using matched blood and stool specimens from screening-guideline eligible subjects.

DETAILED DESCRIPTION:
There is strong evidence supporting the use of FOBT in CRC screening, with the earliest randomized controlled trials demonstrating a reduction in CRC incidence and mortality from CRC screening. Despite the implementation and incremental improvements in gFOBT- and FIT-based tests, they continue to represent a small percentage of CRC screening and currently remain largely the province of large, integrated healthcare delivery systems. Reasons for the limited adoption of stool-based testing are complicated, but include lack of physician recommendation, patient preferences, and cultural barriers.

Availability of a blood-based test may overcome the adoption challenges presently facing stool-based CRC screening and facilitate better compliance with CRC screening guidelines. However, there are currently no FDA-approved in vitro diagnostic tests for detection of CRC in a blood sample. As such, a high through-put blood-based test with performance characteristics similar to fecal testing could satisfy this clinical need.

This study is designed to prospectively collect matched blood and stool specimens and clinical data from screening guideline-eligible subjects found to have invasive colorectal cancer (CRC) at colonoscopy, i.e. AJCC/UICC stages I, II, III, and IV, with collection of specimens and testing after colonoscopy and from screening guideline-eligible subjects with blood and stool specimens collected before colonoscopy. A completed subject will have a FIT result, an Epi proColon result, and a medical diagnosis/colonoscopy determined clinical status (CRC, non-CRC). Demographic and baseline covariates will be reported for each individual.

ELIGIBILITY:
Inclusion Criteria:

Group A

* Willing and able to sign an informed consent and adhere to study requirements
* 50 - 84 years of age at blood and stool sampling
* Colonoscopic diagnosis of colorectal carcinoma
* Colonoscopy within 6 months before inclusion into study
* Blood and stool sampling a minimum of 10 days after colonoscopy and before resection surgery

Group B

* Willing and able to sign an informed consent and adhere to study requirements
* 50 - 84 years of age at blood and stool sampling
* Able to provide blood and stool sample prior to bowel prep and colonoscopy

Exclusion Criteria:

Group A

* Subject with curative biopsy during colonoscopy

Group A and B

* Previous personal history of CRC or previous colonocopy resulting in a recommendation to repeat colonoscopy at an interval less than 10 years
* Neoadjuvant treatment
* Familial risk for colorectal cancer
* History of inflammatory bowel disease
* Acute or chronic gastritis
* Current diagnosis of any other cancer
* Overt rectal bleeding or bleeding hemorrhoids
* Known infection with HIV, HBV, or HCV
* Subject concurrently receiving intravenous fluid at the time of the sample collection

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from gastroenterology clinics and surgical centers in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of Epi proColon test result compared to FIT result using a 95% confidence interval for difference in sensitivities and differences in specificities below a strictly defined margin. | At completion of testing.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Beck, MD, Principal Investigator — Epigenomics, Inc; Neil Mucci, Study Director — Epigenomics, Inc
Locations (70):
- United States (69):
  - Achieve Clinical Research LLC, Birmingham, Alabama
  - Greater Arizona Gastroenterology Associates, Casa Grande, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - South Orange County Surgical Medical Group, Laguna Hills, California
  - Healthcare Partners Medical Group, Los Angeles, California
  - Futura Research, Inc., Montebello, California
  - Southern California Research Institute Medical Group, Inc., Murrieta, California
  - West Gastroenterology Medical Group, Murrieta, California
  - Diverse Research Solutions, LLC, Oxnard, California
  - Inland Gastroenterology Medical Associates, Inc., Redlands, California
  - Santa Monica Research Institute, Santa Monica, California
  - Innovative Clinical Research Institute, Whittier, California
  - Gastroenterology Associates of Fairfield County, Bridgeport, Connecticut
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Zasa Clinical Research, Boyton Beach, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Center for Gastrointestinal Disorders, Hollywood, Florida
  - Palm Springs Research Institute, Inc, Miami, Florida
  - United Clinical Research, Corp., Miami, Florida
  - Advance Medical Research Service Corp., Miami, Florida
  - Physicians Regional Medical Center, Naples, Florida
  - Advance Medical Research Group, Palm Harbor, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - PMI Research, Atlanta, Georgia
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Saint Francis Cancer Care Center, Indianapolis, Indiana
  - Trover Center for Clinical Studies, Madisonville, Kentucky
  - New Orleans Research Institute, Metairie, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Commonwealth Clinical Trials, Brockton, Massachusetts
  - Detroit Clinical Research Center, Novi, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Troy Gastroenterology PC Center for Digestive Health, Troy, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Binghampton Gastroenterology Associates, Binghampton, New York
  - Life Medi-research and Management, Brooklyn, New York
  - Bassett Healthcare Center, Cooperstown, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - New York Gastroenterology Associates, LLP, New York, New York
  - Montefiore - Einstein Cancer Care Center, New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Atlantic Medical Group, Kinston, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Piedmont Medical Research Associates, LLC, Winston-Salem, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - Lillestol Research, LLC, Fargo, North Dakota
  - Gastroenterology Research Consultants of Greater Cincinnati, Cincinnati, Ohio
  - Bend Memorial Clinic, Bend, Oregon
  - Clinical Trials of America, Inc., Eugene, Oregon
  - Bux-Mont Gastroenterology Associates, Sellersville, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Gastroenterology Associates, Kingsport, Tennessee
  - Independent Clinical Research, LLC, Carrolton, Texas
  - Digestive Associates of Houston, Spring, Texas
  - Spring Gastroenterology, Spring, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Multicare Health Systems, Medical Oncology, Tacoma, Washington
  - Dean Foundation Medical Research, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin
- Clinical Research of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Johnson DA, Barclay RL, Mergener K, Weiss G, Konig T, Beck J, Potter NT. Plasma Septin9 versus fecal immunochemical testing for colorectal cancer screening: a prospective multicenter study. PLoS One. 2014 Jun 5;9(6):e98238. doi: 10.1371/journal.pone.0098238. eCollection 2014. PMID 24901436